CLINICAL TRIAL: NCT00924950
Title: An Open-Label, Bilaterally-Controlled Single Center Study to Compare the Efficacy of Taclonex Ointment With Hydrogel Patch Occlusion to Taclonex Ointment Without Occlusion in the Treatment of Plaque-Type Psoriasis
Brief Title: Taclonex Ointment With Hydrogel Patch Occlusion for the Treatment of Psoriasis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H5939-31328-02
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2012-12-05 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Plaque Psoriasis; Psoriasis Vulgaris
Keywords: Psoriasis; Plaque psoriasis, with bilateral symmetrical lesions.; A diagnosis of stable plaque-type psoriasis vulgaris; with at least one pair of symmetric lesions on either; the trunk, arms, or legs that would serve as target lesions.
MeSH Terms: conditions — Psoriasis; Rhabdomyosarcoma, Alveolar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taclonex Ointment/Hydrogel Patch Applied Topically Once Daily (Active Comparator): Taclonex ointment once daily used to treat one psoriatic plaque, along with the Hydrogel Patch used once daily.
  Interventions: Drug: Taclonex Ointment and Hydrogel Patch
- Taclonex Ointment Topically Once Daily (Active Comparator)
  Interventions: Drug: Taclonex Ointment

INTERVENTIONS:
Drug: Taclonex Ointment and Hydrogel Patch — Each patient will have bilateral symmetrical psoriatic plaques. One plaque will be treated with Taclonex Ointment daily along with Hydrogel Patch daily. All treatment will be for 4 weeks.
  Arms: Taclonex Ointment/Hydrogel Patch Applied Topically Once Daily
Drug: Taclonex Ointment — Taclonex ointment daily for one psoriatic plaque.
  Arms: Taclonex Ointment Topically Once Daily

SUMMARY:
The purpose of this study is to determine whether using Taclonex ointment under a hydrogel patch is more effective than using the ointment alone in treating psoriasis. Taclonex ointment is currently FDA approved for use on psoriasis. The hydrogel patch is a type of adhesive pad and contains no medications. It is currently FDA approved and has been shown to be safe and virtually free of side effects. The hypothesis is that psoriatic plaques which are treated with Taclonex ointment under a hydrogel patch will be more effectively treated compared to psoriatic plaques treated with Taclonex alone.

DETAILED DESCRIPTION:
This will be an open label, bilaterally-controlled single center study. Thirty subjects with plaque type psoriasis will be enrolled in the study. All subjects will receive treatment on two target lesions that are similar in erythema, scaling and induration, and symmetric in anatomic location. The severity of their target lesions will be assessed using a modified Psoriasis Area and Severity Index (PASI) scoring system (Appendix A). Symmetrical target lesions must each be rated at a PASI score equal to or greater than 7 and be within 1 PASI score of each other.

All subjects will apply Taclonex ointment to both target lesions once daily for 4 weeks. The occlusive dressing will be applied by the subject to one of the two symmetrical target lesions once daily for 4 weeks. The occlusive dressing will be removed by the patient if he/she experiences warmth, irritation, increased erythema, and/or itching. If the patch is removed due to these symptoms and signs, the subject will leave the lesion un-occluded until for 24 hours, at which time a new occlusive dressing will be placed.

After the initial 4 weeks of treatment, there will be a follow up period of 6 weeks during which no treatment is used.

Subjects will be restricted from using systemic therapies for psoriasis during this study, including Psoralen Ultraviolet A (PUVA) photochemotherapy and herbal therapies. All topical medications, except the study medications, and UVB phototherapy are prohibited on the target lesions. All of the other psoriasis lesions on the body can be treated as usual with other topical medications and Ultraviolet B (UVB) phototherapy as long as it does not impact on the two target lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed the informed consent form and Health Information Portability and Accountability Act (HIPAA) authorization form;
2. Male or female subject at least 18 years of age;
3. A diagnosis of stable plaque-type psoriasis vulgaris with at least one pair of symmetric lesions on either the trunk, arms, or legs that would serve as target lesions. Paired target lesions must be in similar anatomic locations (e.g., right and left elbows or right and left knees) and have roughly equivalent (no more than one point difference) modified Psoriasis Area Severity Index (PASI) scores. Each paired target lesions must have PASI scores equal to or greater than 7;
4. Any additional diagnoses must, in the investigator's opinion, not preclude the subject from safely participating in this study or interfere with the evaluation of the subject's psoriasis;
5. Psoriasis must be clinically stable for at least 30 days before enrollment;
6. Subject is able to discontinue the use of any medication or therapy for relief of psoriasis in the target areas to be treated;
7. Subject is able to discontinue the use of any systemic medication or therapy (e.g. oral or injectable psoriasis medications, PUVA photochemotherapy, herbal remedies, etc.) for psoriasis;
8. Subject must be reliable and mentally competent to complete study measurements;
9. Subject is able to understand and agrees to comply with study requirements, attend study visits, and comply with the restrictions during the study.

Exclusion Criteria:

1. Subject has a skin disorder other than psoriasis in the target areas to be evaluated;
2. Known hypersensitivity to any component of the test medications;
3. Pigmentation, extensive scarring, or pigmented lesions in affected areas that would interfere with evaluation of efficacy parameters;
4. Clinically infected psoriasis at baseline;
5. Guttate, pustular, erythrodermic, or other non-plaque forms of psoriasis;
6. Spontaneously worsening or improving psoriasis within 30 days of enrollment;
7. Any evidence of atrophy in the areas selected for treatment with topical corticosteroid;
8. Topical or intralesional therapies (other than emollients) or UVB phototherapy on potential target lesions within two weeks of starting study treatment;
9. Systemic therapy, PUVA phototherapy, or a systemic investigational therapy for psoriasis within 30 days prior to study entry;
10. Treatment with topical investigational therapy of the target lesions within 30 days prior to study entry;
11. Subject is considered unreliable as to medication compliance or adherence to scheduled appointments as determined by the investigators.
12. Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis Skin and Treatment Center, San Francisco, California, United States

REFERENCES:
- [Background] Griffiths CE, Tranfaglia MG, Kang S. Prolonged occlusion in the treatment of psoriasis: a clinical and immunohistologic study. J Am Acad Dermatol. 1995 Apr;32(4):618-22. doi: 10.1016/0190-9622(95)90347-x. PMID 7534777
- [Background] Fenton C, Plosker GL. Calcipotriol/betamethasone dipropionate: a review of its use in the treatment of psoriasis vulgaris. Am J Clin Dermatol. 2004;5(6):463-78. doi: 10.2165/00128071-200405060-00012. PMID 15663344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at the University of California at San Francisco (UCSF) Psoriasis and Skin Treatment Center.
Pre-assignment Details: Patients were assessed for psoriasis severity as well as washout from other concomitant medications
Groups:
- Ointment + Patch vs. Ointment Alone: Taclonex (calcipotriene 0.005% and betamethasone dipropionate 0.064%) ointment used topically to treat one psoriatic plaque with Hydrogel patch used over for occlusion for 6-8 hours daily. Within the same patient another patch of similar severity was chosen and was treated with Taclonex ointment alone without hydrogel patch occlusion
Period: Overall Study
Arm/Group | Ointment + Patch vs. Ointment Alone
Started | 30
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ointment + Patch vs. Ointment Alone
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Gender was not measured in each arm
  Male | NA — Gender was not measured in each arm
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Modified PASI Score at Week 4 Compared to Baseline
Description: Modified psoriasis severity index measures erythema, induration, and scaling each measured from 0-4, with a maximum summed score of 12. A higher score means greater psoriasis severity and a lower score means lower psoriasis severity.
Time Frame: 4 weeks
Population: The number of participants was chosen by our budget restrictions. 35 patients were enrolled. 5 patients were lost to follow-up.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Groups:
- Taclonex Ointment Occluded With Hydrogel Patch: Taclonex (calcipotriene 0.005% and betamethasone dipropionate 0.064%) ointment used daily topically to treat one psoriatic plaque, occluded with hydrogel patch for 6-8 hours each day.
- Taclonex Alone: Taclonex (calcipotriene 0.005% and betamethasone dipropionate 0.064%) ointment used daily without hydrogel patch.
Arm/Group | Taclonex Ointment Occluded With Hydrogel Patch | Taclonex Alone
Number analyzed (Participants) | 30 | 30
Units on a scale | 0.86 [0.40 to 1.31] | 2.2 [1.7 to 3.58]
Statistical Analysis 1: Comparison: Taclonex Ointment Occluded With Hydrogel Patch vs Taclonex Alone; Test type: Superiority; p = 0.0008, t-test, 2 sided; Mean Difference (Final Values) = 0.8571

2. Secondary Outcome: Change in Modified PASI Scores Between Week 4 and Week 6 During the Follow-up Period. This is to Determine Whether There is Further Improvement of Psoriasis After the Cessation of Occlusion
Description: Change in Modified PASI Scores Between Week 4 and Week 6 During the Follow-up Period. This is to Determine Whether There is Further Improvement of Psoriasis After the Cessation of Occlusion.
Time Frame: 6 Weeks
Population: This outcome measure was not analyzed due to termination of the study
Arm/Group | Taclonex Ointment/Hydrogel Patch Applied Topically Once Daily | Taclonex Ointment Topically Once Daily
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ointment + Patch vs. Ointment Alone
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No